CLINICAL TRIAL: NCT00702273
Title: Follow-up Protocol to Collect the Outcome of Frozen-thawed Embryo Transfer Cycles After Cryopreservation of Embryos in Clinical Trial 38819
Brief Title: Follow-up Study of Frozen-thawed Embryo Transfer (FTET) Cycles After Cryopreservation of Embryos in Clinical Trial P05787 (P05716)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05716; 2004-004773-28 (EudraCT Number); 38831 (Other: Organon); MK-8962-009 (Other: Merck)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2022-02

CONDITIONS: In Vitro Fertilization
Keywords: In-vitro fertilization; Controlled Ovarian Stimulation; Cumulative pregnancy data; Follow-up
MeSH Terms: interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta; ganirelix; Progesterone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 150 µg Corifollitropin Alfa: Participants from the base study P05787 (NCT00696800), received a single subcutaneous (SC) injection of 150 µg Corifollitropin Alfa (Org 36286) on menstrual cycle Day 2/3 (Day 1); 7 daily SC injections from Days 1 to 7 with placebo-recombinant Follicle Stimulating Hormone (recFSH); followed by daily SC injections with 200 IU recFSH up to the day of human chorionogonadotropin (hCG). Daily SC injections of Ganirelix were given from Day 5 to the day of hCG; at which time a single dose of hCG was given when 3 follicles >= 17 mm. On the day of oocyte pick up (OPU) daily doses of progesterone were started, for up to 6 weeks or menses. Eligible participants from the base study were enrolled in follow up study P05716, where no study treatments were given, and embryos obtained in the base study underwent FTET cycles.
  Interventions: Drug: 150 µg Corifollitropin Alfa; Drug: Placebo for RecFSH/Follitropin beta; Biological: 200 IU RecFSH/Follitropin beta (Days 8 to hCG); Drug: Ganirelix; Biological: hCG; Biological: Progesterone
- 200 IU RecFSH: Participants from the base study P05787 (NCT00696800), received a single SC injection of placebo Corifollitropin Alfa on menstrual cycle day 2/3 (Day 1); 7 daily SC injections with 200 IU recFSH from Days 1 to 7; followed by daily SC injections with 200 IU recFSH up to the day of hCG. Multiple daily SC injections of Ganirelix were given from Day 5 to the day of hCG; at which time a single dose of hCG was given when 3 follicles >= 17 mm. On the day of OPU daily doses of progesterone were started and continued for up to 6 weeks or menses. Eligible participants from the base study were enrolled in follow up study P05716, where no study treatments were given, and embryos obtained in the base study underwent FTET cycles.
  Interventions: Biological: 200 IU RecFSH/Follitropin beta (Days 1 to 7); Drug: Placebo for Corifollitropin Alfa; Biological: 200 IU RecFSH/Follitropin beta (Days 8 to hCG); Drug: Ganirelix; Biological: hCG; Biological: Progesterone

INTERVENTIONS:
Drug: 150 µg Corifollitropin Alfa — On the morning of day 2 or 3 of the menstrual cycle (Stimulation Day 1), a single SC injection of 150 μg (0.5 mL) Corifollitropin Alfa was administered in the abdominal wall.
  Groups: 150 µg Corifollitropin Alfa
Biological: 200 IU RecFSH/Follitropin beta (Days 1 to 7) — Daily SC injections with 200 IU fixed dose recFSH were started on Stimulation Day 1 and continued up to and including Stimulation Day 7.
  Groups: 200 IU RecFSH
Drug: Placebo for Corifollitropin Alfa — Pre-filled syringe containing an identical solution when compared to Corifollitropin Alfa. On the morning of day 2 or 3 of the menstrual cycle (Stimulation Day 1), a single SC injection was administered in the abdominal wall.
  Groups: 200 IU RecFSH
Drug: Placebo for RecFSH/Follitropin beta — Identical ready-for-use solution, but without the active ingredient, supplied in cartridges for SC injection with the Follistim Pen. Daily SC injections were started on Stimulation Day 1 and continued up to and including Stimulation Day 7.
  Groups: 150 µg Corifollitropin Alfa
Biological: 200 IU RecFSH/Follitropin beta (Days 8 to hCG) — From Stimulation Day 8 onwards a daily SC dose of 200 IU recFSH was administered up to and including the Day of hCG.
Drug: Ganirelix — On Stimulation Day 5 a daily SC injection of 0.25 mg was started, which continued up to and including the day of hCG
Biological: hCG — When 3 follicles >= 17 mm were observed by USS, a single dose of 10,000 IU/USP hCG was administered; or, for those at risk for Ovarian Hyperstimulation Syndrome (OHSS), a lower dose of 5,000 IU/USP
Biological: Progesterone — On the day of OPU, luteal phase support was started by administering micronized progesterone of at least 600 mg/day vaginally, or at least 50 mg/day intramuscular (IM), which continued for at least 6 weeks, or up to menses.

SUMMARY:
To collect the outcome of frozen-thawed embryo transfer cycles after the embryos are cryopreserved up to at least 1 year in Trial P05787 (NCT00696800), in order to estimate the cumulative pregnancy rate for each treatment group.

DETAILED DESCRIPTION:
This is a follow-up protocol to collect the outcome of frozen-thawed embryo transfer cycles, performed after the embryos are cryopreserved up to at least 1 year in Trial P05787 (NCT00696800), to enable estimation of the cumulative pregnancy rate for each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Participants from whom embryos have been cryopreserved in Base Trial P05787 (NCT00696800), of which at least one embryo is thawed for use in a subsequent FTET cycle;
* Able and willing to give informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women from whom embryos have been cryopreserved in Base Trial P05787 (NCT00696800).
Sampling Method: Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2006-04-19 (Actual); Primary Completion 2009-05-19 (Actual); Study Completion 2009-05-31 (Actual)

REFERENCES:
- [Derived] Boostanfar R, Mannaerts B, Pang S, Fernandez-Sanchez M, Witjes H, Devroey P; Engage Investigators. A comparison of live birth rates and cumulative ongoing pregnancy rates between Europe and North America after ovarian stimulation with corifollitropin alfa or recombinant follicle-stimulating hormone. Fertil Steril. 2012 Jun;97(6):1351-8. doi: 10.1016/j.fertnstert.2012.02.038. Epub 2012 Mar 28. PMID 22459628

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period one consists of participants from the base study P05787 (NCT00696800), randomized to treatment groups Corifollitropin Alfa (Cori Alfa) (Org 36286) or recombinant Follicle Stimulating Hormone (recFSH). Period two consists of eligible participants (N = 344) from the base study who enrolled in the follow up study P05716.
Groups:
- 150 µg Corifollitropin Alfa: Participants from the base study P05787 (NCT00696800), received a single subcutaneous (SC) injection of 150 µg Corifollitropin Alfa on menstrual cycle Day 2/3 (Day 1); 7 daily SC injections from Days 1 to 7 with placebo-recFSH); followed by daily SC injections with 200 IU recFSH up to the day of human chorionogonadotropin (hCG). Daily SC injections of Ganirelix were given from Day 5 to the day of hCG; at which time a single dose of hCG was given when 3 follicles >= 17 mm. On the day of oocyte pick up (OPU) daily doses of progesterone were started, for up to 6 weeks or menses. Eligible participants from the base study were enrolled in follow up study P05716, where no study treatments were given, and embryos obtained in the base study underwent frozen thawed embryo transfer (FTET) cycles.
Period: Base Study P05787 (NCT00696800)
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH
Started | 757 (Participants randomized to the base study P05787 (NCT00696800)) | 752 (Participants randomized to the base study P05787 (NCT00696800))
Treated | 756 (Participants from the Intent to Treat group (ITT) from the base study P05787 (NCT00696800)) | 750 (Participants from the Intent to Treat group (ITT) from the base study P05787 (NCT00696800))
Completed | 672 (To complete study, participants from the base study P05787 (NCT00696800) had embryos transferred) | 704 (To complete study, participants from the base study P05787 (NCT00696800) had embryos transferred)
Not Completed | 85 | 48
Period: Follow Up Study P05716 (NCT00702273)
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH
Started | 168 (Participants from base study,who had at least one embryo thawed for a FTET cycle.) | 176 (Participants from base study, who had at least one embryo thawed for a FTET cycle)
Completed | 148 (Participants with embryo transfer in any FTET cycle) | 147 (Participants with embryo transfer in any FTET cycle)
Not Completed | 20 | 29

BASELINE CHARACTERISTICS:
Population: Eligible participants from base study P05787 (NCT00696800) who enrolled in follow up study P05716
Groups:
- 150 µg Corifollitropin Alfa: Participants from the base study P05787 (NCT00696800), received a single subcutaneous (SC) injection of 150 µg Corifollitropin Alfa on menstrual cycle Day 2/3 (Day 1); 7 daily SC injections from Days 1 to 7 with placebo-recFSH); followed by daily SC injections with 200 IU recFSH up to the day of human chorionogonadotropin (hCG). Daily SC injections of Ganirelix were given from Day 5 to the day of hCG; at which time a single dose of hCG was given when 3 follicles >= 17 mm. On the day of oocyte pick up (OPU) daily doses of progesterone were started, for up to 6 weeks or menses. Eligible participants from the base study were enrolled in follow up study P05716, where no study treatments were given, and embryos obtained in the base study underwent FTET cycles.
- Total: Total of all reporting groups
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH | Total
Number analyzed (Participants) | 168 | 176 | 344
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.1 (3.8) | 31.3 (3.0) | 31.2 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 176 | 344
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Ongoing Pregnancy (Cumulative Ongoing Pregnancy Rate)
Description: An ongoing pregnancy is the presence of at least one fetus with heart activity at least 10 weeks after embryo transfer or confirmed by live birth.The cumulative ongoing pregnancy rate is 100 times the number of participants with an ongoing pregnancy either immediately after embryo transfer in base Trial P05787 (NCT00696800), or after one or more FTET cycles in follow-up Trial P05716 following cryopreservation, divided by the total number of participants that started treatment in base Trial P05787 (NCT00696800). Participants who did not have cryopreserved embryos, or embryo transfers in the FTET cycle(s), were considered 'not pregnant'.
Time Frame: Up to 1 year after embryo transfer in base trial P05787 (NCT00696800), and FTET cycles in follow up trial
Population: ITT group from base trial P05787, consisting of randomized participants who were treated with Corifollitropin Alfa or recFSH.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH
Number analyzed (Participants) | 756 | 750
Percentage of participants | 47.2 | 44.9
Statistical Analysis 1: Comparison: 150 µg Corifollitropin Alfa vs 200 IU RecFSH; Treatment groups were compared with a generalized linear model including covariates treatment group, age class and region; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of -8%; Risk Difference (RD) = 2.4, 95% CI 2-sided [-2.6 to 7.4]

2. Secondary Outcome: Percentage of Participants in Follow up Trial With a Miscarriage Per Clinical Pregnancy
Description: Miscarriages were calculated per clinical pregnancy, meaning the presence of at least one gestational sac or confirmed by live birth.
Time Frame: After one or more FTET cycles, up to day of miscarriage (up to 1 year)
Population: Participants enrolled in P05716 Follow Up study that had a clinical pregnancy.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH
Number analyzed (Participants) | 73 | 68
Percentage of participants | 8.2 | 17.6

3. Secondary Outcome: Percentage of Participants in Follow up Trial With a Miscarriage Per Vital Pregnancy
Description: Miscarriages were calculated per vital pregnancy, meaning the presence of at least one fetus with heart activity.
Time Frame: After one or more FTET cycles, up to day of miscarriage (up to 1 year)
Population: Participants enrolled in P05716 Follow Up study that had a vital pregnancy.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH
Number analyzed (Participants) | 67 | 56
Percentage of participants | 0 | 0

4. Secondary Outcome: Percentage of Participants in Follow up Trial With an Ectopic Pregnancy
Description: An ectopic pregnancy is where the embryo implants outside the uterus. Ectopic pregnancies were calculated per total number of participants started in FTET.
Time Frame: After one or more FTET cycles, assessed at least 10 weeks after embryo transfer (up to 1 year)
Population: Participants enrolled in P05716 Follow Up study.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH
Number analyzed (Participants) | 168 | 176
Percentage of participants | 1.2 | 0.6

5. Secondary Outcome: Percentage of Participants in Follow up Trial With a Clinical Pregnancy
Description: A clinical pregnancy is the presence of at least gestational sac or confirmed by live birth. Clinical pregnancies were calculated per attempt, meaning if any stage of in vitro fertilization (IVF) treatment was not achieved, zero values were imputed.
Time Frame: After one or more FTET cycles, assessed at least 10 weeks after embryo transfer (up to 1 year)
Population: Participants enrolled in P05716 Follow Up study, that had an embryo transfer in the respective cycle.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH
Number analyzed (Participants) | 168 | 176
Percentage of participants | 43.5 | 38.6

6. Secondary Outcome: Percentage of Participants in Follow up Trial With a Vital Pregnancy
Description: A vital pregnancy is the presence of at least one fetus with heart activity. Vital pregnancies were calculated per attempt, meaning if any stage of IVF treatment was not achieved, zero values were imputed.
Time Frame: After one or more FTET cycles, assessed at least 10 weeks after embryo transfer (up to 1 year)
Population: Participants enrolled in P05716 Follow Up study, that had an embryo transfer in the respective cycle.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH
Number analyzed (Participants) | 168 | 176
Percentage of participants | 39.9 | 31.8

7. Secondary Outcome: Percentage of Participants in Follow up Trial With an Ongoing Pregnancy
Description: An ongoing pregnancy is the presence of at least one fetus with heart activity at least 10 weeks after embryo transfer or confirmed at live birth. Ongoing pregnancies were calculated per attempt, meaning if any stage of IVF treatment was not achieved, zero values were imputed.
Time Frame: After one or more FTET, assessed at least 10 weeks after embryo transfer or at live birth (up to 1 year)
Population: Participants enrolled in P05716 Follow Up study, that had an embryo transfer in the respective cycle.
Measure: Number; unit: Percentage of participants
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH
Number analyzed (Participants) | 168 | 176
Percentage of participants | 38.7 | 30.7

ADVERSE EVENTS:
Description: Participants who enrolled in Trial P05716 Follow Up. Trial P05716 did not systematically collect Serious Adverse Events (SAEs) or AEs. Instead any reported AEs were unsolicited and non-systematically assessed. Ectopic pregnancies in Outcome Measure 4 were collected as an efficacy rather than a safety endpoint; and were therefore not counted as AEs.
Arm/Group | 150 µg Corifollitropin Alfa | 200 IU RecFSH
Serious Adverse Events (participants affected / at risk) | 1/168 | 0/176
Other Adverse Events (participants affected / at risk) | 0/168 | 0/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 µg Corifollitropin Alfa (N=168) | 200 IU RecFSH (N=176)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning the clinical trial will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably. The Sponsor shall have the right to make its consent conditional upon proper representation of the interpretation of both the Sponsor and the investigator(s) in the discussion of the data in such communications.